CLINICAL TRIAL: NCT05907525
Title: Effect of Sevoflurane and Remimazolam on Arterial Oxygenation During One-lung Ventilation: a Prospective Randomized Controlled Study
Brief Title: Effect of Sevoflurane and Remimazolam on Arterial Oxygenation During One-lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Kim Hee Young, Assistant professor for fund, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 05-2023-133
Record Dates: First submitted 2023-06-05; First posted 2023-06-18 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: One-Lung Ventilation; Thoracic Surgery, Video-Assisted; Remimazolam
Keywords: remimazolam; one-lung ventilation; arterial oxygenation; hypoxic pulmonary vasoconstriction; sevoflurane; thoracic surgery
MeSH Terms: interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam group (Experimental): To induce anesthesia, remimazolam is continuously infused in a dose of 6mg/kg/hr with remifentanil (Ce of 1-4ng/ml) by target-controlled infusion (TCI). Maintenance dose of remimazolam is 1mg/kg/hr, up to 2mg/kg/hr, and remifentanil is titrated to maintain the bispectral index (BIS) between 40 and 60 to achieve appropriate anesthetic depth during general anesthesia.
  Interventions: Drug: Remimazolam
- Sevoflurane group (Active Comparator): To induce anesthesia, 1% propofol 1.5-2.5mg/kg is used with remifentanil (Ce of 1-4ng/ml) by target-controlled infusion (TCI). After patient loses consciousness, anesthesia is maintained through the inhalation of sevoflurane between 1-2 minimum alveolar concentrations (MAC). Remifentanil is titrated to maintain the bispectral index (BIS) between 40 and 60 to achieve appropriate anesthetic depth during general anesthesia.
  Interventions: Drug: 1% propofol

INTERVENTIONS:
Drug: Remimazolam — To induce anesthesia, remimazolam is continuously infused in a dose of 6mg/kg/hr with remifentanil (Ce of 1-4ng/ml) by target-controlled infusion (TCI). Maintenance dose of remimazolam is 1mg/kg/hr, up to 2mg/kg/hr, and remifentanil is titrated to maintain the bispectral index (BIS) between 40 and 60 to achieve appropriate anesthetic depth during general anesthesia.
  Inspired oxygen fraction (FiO2) 1.0 is used during mask ventilation and tracheal intubation. During two lung ventilation (TLV), tidal volumes (8mL/kg predicted body weight), positive end-expiratory pressure (PEEP) 5cmH2O with FiO2 0.3 is applied. At the start of one lung ventilation(OLV), tidal volumes (5mL/kg predicted body weight), PEEP 5cmH2O with FiO2 0.8 is applied. Intraoperative ventilatory frequency is 12 breaths/min, subsequently adjusted to maintain end tidal CO2(ETCO2) ranged between 35-40mmHg.
  Other Names: Byfavo
  Arms: Remimazolam group
Drug: 1% propofol — To induce anesthesia, 1% propofol 1.5-2.5mg/kg is used with remifentanil (Ce of 1-4ng/ml) by target-controlled infusion (TCI). After patient loses consciousness, anesthesia is maintained through the inhalation of sevoflurane between 1-2 minimum alveolar concentrations (MAC), and remifentanil is titrated to maintain the bispectral index (BIS) between 40 and 60 to achieve appropriate anesthetic depth during general anesthesia.
  Inspired oxygen fraction (FiO2) 1.0 is used during mask ventilation and tracheal intubation. During two lung ventilation (TLV), tidal volumes (8mL/kg predicted body weight), positive end-expiratory pressure (PEEP) 5cmH2O with FiO2 0.3 is applied. At the start of one lung ventilation(OLV), tidal volumes (5mL/kg predicted body weight), PEEP 5cmH2O with FiO2 0.8 is applied. Intraoperative ventilatory frequency is 12 breaths/min, subsequently adjusted to maintain end tidal CO2(ETCO2) ranged between 35-40mmHg.
  Other Names: Fresofol MCT 1%
  Arms: Sevoflurane group

SUMMARY:
The goal of this clinical trial is to compare the effect of sevoflurane and remimazolam on arterial oxygenation during one lung ventilation in patients undergoing video-assisted thoracoscopic surgery.

DETAILED DESCRIPTION:
One lung ventilation (OLV) is a mechanical ventilation method used during thoracic surgery to collapse the non-ventilated lung and secure the surgical field. During one lung ventilation, the pulmonary artery of the collapsed lung undergoes vasoconstriction in response to hypoxia, which increases the blood flow of the normally ventilated lung as a compensatory physiological response. This is known as hypoxic pulmonary vasoconstriction (HPV). Therefore, by using HPV, arterial blood oxygenation can be maintained and pulmonary shunting can be reduced, preventing hypoxemia during one lung ventilation.

The two most commonly used anesthetics in thoracic surgery are sevoflurane, an inhaled anesthetic, and propofol, an intravenous anesthetic. Previous studies have shown that there were no significant differences between two anesthetics on arterial oxygenation during one lung ventilation because sevoflurane administered in clinical concentrations of 1 minimum alveolar concentration (MAC) resulted in similar changes in shunt fraction as did propofol.

However, the effect of remimazolam on arterial blood oxygenation and intrapulmonary shunt during one lung ventilation has not been revealed. Therefore, this study is designed to compare the effect of remimazolam and sevoflurane anesthesia on arterial oxygenation during one lung ventilation in patients undergoing video-assisted thoracoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing video-assisted thoracoscopic surgery
* 19 years of age or older, less than 80 years old
* The American Society of Anesthesiologists (ASA) classification I-Ⅲ physical status

Exclusion Criteria:

* Patients with known allergy to benzodiazepine, propofol
* Patients with galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
* Patients with hypersensitivity to Dextran40
* Patients with end stage renal disease requiring hemodialysis
* Patients with history of acute angle glaucoma
* Emergency operation
* Patients with unstable hemodynamics requiring inotropics
* Patients with preoperative oxygen supplement
* Preoperative forced expiratory volume (FEV1) less than 40% of predicted
* Preoperative ejection fraction less than 50%

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
PaO2 after 30 minutes of OLV (T2) | arterial blood sampling will be taken over four times: T0 (after 10 minute of TLV in lateral decubitus position), T1 (after 15 minutes of OLV), T2 (after 30 minutes of OLV), T3 (after 60 minutes of OLV)
  compare the arterial oxygenation after 30 minutes of one lung ventilation between two groups

SECONDARY OUTCOMES:
Changes of PaO2 | During 60 minutes of OLV
  Compare the changes of PaO2 between two groups.
Changes of PaCO2 | During 60 minutes of OLV
  Compare the changes of PaCO2 between two groups.
Changes of P/F ratio | During 60 minutes of OLV
  Compare the changes of PaO2/FiO2 ratio between two groups.
The lowest PaO2 | During 60 minutes of OLV
  Compare the lowest PaO2 between two groups.
Changes of ORI | During 60 minutes of OLV
  Compare the changes of oxygen reserve index between two groups.
Changes of MAP | During 60 minutes of OLV
  Compare the changes of mean arterial pressure between two groups.

OTHER OUTCOMES:
cardiac output | During 60 minutes of OLV
  Compare the cardiac output using Masimo LiDCO™ hemodynamic monitoring system
airway pressure | During 60 minutes of OLV
  Compare the peak airway pressure between two groups

CONTACTS AND LOCATIONS:
Overall Officials: Hee Young Kim, MD. PhD, Study Chair — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Please Select, South Korea

IPD SHARING:
Plan to Share IPD: No